CLINICAL TRIAL: NCT03674385
Title: Evaluation of the Clinical Outcome of Vitamin E as Adjuvant Therapy in Patients With Clomiphene Citrate Resistant Polycystic Ovary Syndrome
Brief Title: Efficacy of Vit E in PCOS Resistant to Clomiphene Citrate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, Ahmed Abbas Morsy Morsy, pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL 191
Record Dates: First submitted 2018-08-15; First posted 2018-09-17 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Clomiphene Citrate Resistant Polycystic Ovary Syndrome
Keywords: Vitamin E; Polycystic ovary
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Vitamin E; Metformin; Clomiphene

STUDY DESIGN:
Intervention Model Description: prospective randomized controlled open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin E group (Experimental): 30 patient
  Interventions: Dietary Supplement: vitamin E; Drug: Metformin; Drug: Clomiphene Citrate
- control group (Active Comparator): clomiphene
  Interventions: Drug: Metformin; Drug: Clomiphene Citrate

INTERVENTIONS:
Dietary Supplement: vitamin E — Vitamin E is sold as a dietary supplement, either by itself or incorporated into a multivitamin product. it also has anti-oxidant effect
  Other Names: toco 1000
  Arms: vitamin E group
Drug: Metformin — Metformin is in the biguanide class. It works by decreasing glucose production by the liver and increasing the insulin sensitivity of body tissues. It is also used in the treatment of polycystic ovary syndrome (PCOS)
  Other Names: cidophage
Drug: Clomiphene Citrate — is a medication used to treat infertility in women who do not ovulate
  Other Names: clomid

SUMMARY:
This study evaluate the addition of Vit E to clomiphene citrate in the treatment of poly cystic ovary.Half the patients will receive both Vit E and clomiphene citrate the other half will receive clomiphene citrate only.

DETAILED DESCRIPTION:
Clomiphene and vit E each used in treatment of pco but they do so by different mechanisms.

Clomifene is in the selective estrogen receptor modulator (SERM) family of medication. It works by causing the release of gonadotropin-releasing hormone by the hypothalamus, and subsequently gonadotropin from the anterior pituitary.

Vit E is used in treatment of pco due its anti-oxidant effect.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be diagnosed as having PCOS according to the Rotterdam criteria for diagnosis of PCOS
2. Age between 18 and 39 years.
3. Period of infertility >1 years.
4. No treatment taken during the last 2 months.
5. Patients who have previously received clomiphene citrate (CC) and being diagnosed as having CC resistance

Exclusion Criteria:

1. History of pelvic surgery or infertility factor other than anovulation
2. Endocrine disorders in the form of hypothyroidism or hyperthyroidism, hyperprolactinemia, and Cushing syndrome, as detected by history, examination, or investigations.
3. Known cases of endometriosis (approved histologically), uterine anomaly or hydrosalpinx, retinitis pigmentosa and vitamin K deficiency.
4. Consumption of vitamin and antioxidant supplementations in the last three-months before the trial start date.
5. Male factor infertility (sperm count < 5 million per milliliter, normal morphology <4%).
6. Elevated serum prolactin, T.S.H and F.S.H.
7. Patients diagnosed with diabetes mellitus

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
ovulation rate | 3 months
  Follicles measure more than 18 mm will be considered mature follicles.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Center of Infertility, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: No